CLINICAL TRIAL: NCT02170844
Title: Safety, Pharmacokinetics and Pharmacodynamics After Single Rising Oral Doses of 50, 150 and 350 mg BIBR 1048 MS as Capsules in Healthy Subjects of Japanese and Caucasian Origin. Double-blind at Each Dose Level, Placebo-controlled, Randomised Study
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics After Single Rising Oral Doses of BIBR 1048 MS as Capsules in Healthy Subjects of Japanese and Caucasian Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.28
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BIBR 1048 MS (Japanese) (Experimental): Japanese subjects received an increasing dose (50 mg to 150 mg) of BIBR 1048 MS
  Interventions: Drug: BIBR 1048 MS
- BIBR 1048 MS Placebo (Japanese) (Placebo Comparator): Japanese subjects will receive placebo of BIBR 1048 MS
  Interventions: Drug: Placebo of BIBR 1048 MS
- BIBR 1048 MS (Caucasian) (Experimental): Caucasian subjects received an increasing dose (50 mg to 150 mg) of BIBR 1048 MS
  Interventions: Drug: BIBR 1048 MS
- BIBR 1048 MS Placebo (Caucasian) (Placebo Comparator): Japanese subjects will receive placebo of BIBR 1048 MS
  Interventions: Drug: Placebo of BIBR 1048 MS

INTERVENTIONS:
Drug: BIBR 1048 MS
  Arms: BIBR 1048 MS (Caucasian); BIBR 1048 MS (Japanese)
Drug: Placebo of BIBR 1048 MS
  Arms: BIBR 1048 MS Placebo (Caucasian); BIBR 1048 MS Placebo (Japanese)

SUMMARY:
To investigate and compare safety, pharmacokinetics and pharmacodynamics of BIBR 1048 MS following oral administration of single rising doses from 50 mg to 350 mg in healthy male subjects of Japanese and Caucasian origin. This was the first administration of this substance to subjects of Japanese origin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR, Respiratory Rate and tympanic body temperature), 12- lead ECG, clinical laboratory tests
   * 1.1. No finding deviating from normal and of clinical relevance
   * 1.2. No evidence of a clinically relevant concomitant disease
2. Age ≥20 and Age ≤45 years
3. BMI ≥18 and BMI ≤25 kg/m2 (Body Mass Index)
4. Japanese subjects were from a well-defined Japanese population, both parents of Japanese origin and the subjects have Japanese passport and had lived ≤ 8 years outside Japan.
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

1. Current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women, or an unwillingness if the male subject to use an adequate form of contraception as well as having their female partner(s) use another form of contraception (if the woman could become pregnant) from the time of the first dose administration until after follow up
3. Current diseases of the central nervous system (such as epilepsy), or psychiatric disorders or neurological disorders
4. History of clinically significant orthostatic hypotension, clinically significant current or past fainting spells or blackouts.
5. Chronic or relevant acute infections
6. History of - allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator

   * any bleeding disorder including prolonged or habitual bleeding
   * other hematologic disease
   * cerebral bleeding (e.g. after a car accident)
   * concussions (head trauma resulting in injuring to brain) with or without loss of consciousness
7. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives, whichever is shorter, of the respective drug prior to administration or during the trial
8. Use of Acetylsalicylic-Acid (ASA)-containing over-the-counter medications, clopidogrel or ticlopidine or dipyridamole, chronic administration of Non Steroidal Antiinflammatory Drugs (NSAIDs) (COX-2 inhibitors excluded), coumadin like anticoagulants, chronic use of corticosteroids, heparin and fibrinolytic agents within 14 days prior to administration or during the trial.
9. Use of all other medication including over the counter (medicinal cream, vitamin, eye drop etc.) within 7 days prior to administration or during the trial.
10. Participation in another trial with an investigational drug within three months prior to administration or during the trial
11. Smoker (> 10 cigarettes/day or > 3 cigars/day or > 3 pipes/day)
12. Inability to refrain from smoking on trial days
13. Alcohol abuse (more than 21unit/week)
14. History of drug abuse
15. Blood donation (more than 100 mL within three months prior to screening administration and any blood donation from screening to follow-up)
16. Excessive physical activities (within one week prior to administration or during the trial and until follow-up)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Known hypersensitivity to the drug or its excipients

    Exclusion criteria specific for this study:
20. History of any familial bleeding disorder
21. Thrombocytes < 150000/micro L

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood pressure (BP) | At screening (day -14 to -3), at day -1, pre-dose, 2, 8, 24, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in pulse rate (PR) | At screening (day -14 to -3), at day -1, pre-dose, 2, 8, 24, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in respiratory rate | At screening (day -14 to -3), at day -1, pre-dose, 2, 8, 24, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in tympanic body temperature | At screening (day -14 to -3), at day -1, pre-dose, 2, 8, 24, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in 12-Lead electrocardiogram (ECG) | At screening (day -14 to -3), at day -1, pre-dose, 2, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in haematology | At screening (day -14 to -3), at day -1 (pre-dose), 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in blood chemistry | At screening (day -14 to -3), at day -1 (pre-dose), 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Change from baseline in urinalysis | At screening (day -14 to -3), at day -1 (pre-dose), 4, 8, 12, 24, 36, 48 h after administration and on visit 5 (day 10 to day 14 after administration)
Occurence of adverse events | Up to visit 5 (day 10 - 14)

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
tmax (time from dosing to maximum concentration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable point) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
λz (terminal rate constant in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
MRTpo (mean residence time of the analyte in the body after po administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
  (Pharmacokinetic parameters)
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36 and 36-48 h after administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36 and 36-48 h after administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36 and 36-48 h after administration
Change from baseline for activated Partial Thromboplastin Time (aPTT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
Change from baseline for Ecarin clotting time (ECT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
  (Pharmacodynamic parameters)
Change from baseline for thrombin time (TT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration
Change from baseline for international normalised ratio (INR) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after administration